CLINICAL TRIAL: NCT00991692
Title: A Multisite Trial of ACQUIREc Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Stephanie C. DeLuca, PhD, UAB
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: deluca-ms1
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Hemiparetic Cerebral Palsy
Keywords: Pediatric CI Therapy; ACQUIREc Therapy; Dosage; Occupational Therapy; Physical Therapy; Cerebral Palsy; Hemiparesis
MeSH Terms: conditions — Cerebral Palsy; Paresis | interventions — Occupational Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment dosage levels examined (Experimental)
  Interventions: Other: Therapy services (ACQUIREc Therapy)

INTERVENTIONS:
Other: Therapy services (ACQUIREc Therapy) — Dosage levels that are associated with the efficacy of intensive therapeutic services provided by OT and PT professionals.
  Other Names: Occupational Therapy; Physical Therapy; Pediatric CI Therapy; ACQUIREc Therapy

SUMMARY:
A multisite trial to testing different dosage levels of a systematic form of Pediatric Constraint-Induced (CI) Therapy called ACQUIREc Therapy. The high dosage treatment involved 6 hours of daily therapy services for 21 days. This was compared to a moderate dosage level of 3 hours of daily therapy services for 21 days. It was hypothesized that children receiving the higher therapy dosage would have greater and more clinically significant benefits from ACQUIREc Therapy but that both groups of children would benefit from the therapy services.

ELIGIBILITY:
Inclusion Criteria:

* Children 3-6 years of age
* Hemiparetic CP

Exclusion Criteria:

* No prior CI therapy treatments
* No Botox for 6-months

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie C DeLuca, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] DeLuca SC, Case-Smith J, Stevenson R, Ramey SL. Constraint-induced movement therapy (CIMT) for young children with cerebral palsy: effects of therapeutic dosage. J Pediatr Rehabil Med. 2012;5(2):133-42. doi: 10.3233/PRM-2012-0206. PMID 22699104